CLINICAL TRIAL: NCT01338415
Title: A Prospective, Multicenter, Open-label Extension of FUTURE 3 to Assess the Safety, Tolerability and Efficacy of the Pediatric Formulation of Bosentan Two Versus Three Times a Day in Children With Pulmonary Arterial Hypertension
Brief Title: FUTURE 3 Study Extension
Acronym: FUTURE 3 Ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-374; 2010-021793-12 (EudraCT Number)
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pediatric; pulmonary arterial hypertension; bosentan; Tracleer
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan

ARMS (2):
- bosentan 2mg/kg b.i.d. (Experimental): Patients who received 2 mg/kg bosentan twcie daily (b.i.d.) during the FUTURE 3 core study and continued with the same dose regimen during the extension study
  Interventions: Drug: Bosentan
- bosentan 2mg/kg t.i.d. (Experimental): Patients who received 2 mg/kg bosentan 3 times a day (t.i.d.) during the FUTURE 3 core study and continued with the same dose regimen during the extension study
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — Oral dispersible tablet administered as 2mg/kg two (b.i.d.) or three (t.i.d.) times per day
  Other Names: ACT-050088

SUMMARY:
The objectives of the FUTURE 3 Study Extension are to evaluate the long-term safety, tolerability and efficacy of the pediatric formulation of bosentan two versus three times a day in children with Pulmonary Arterial Hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who completed the FUTURE 3 core study (AC-052-373) or prematurely discontinued due to PAH-progression, if bosentan was not permanently discontinued
2. Patients who tolerated bosentan pediatric formulation and for whom bosentan is considered beneficial at the end of the FUTURE 3 core study (AC-052-373)
3. Signed informed consent by the parents or the legal representatives prior to any study-mandated procedure.

Exclusion Criteria:

1. Known intolerance or hypersensitivity to bosentan or any of the excipients of the dispersible bosentan tablet
2. Any clinically significant laboratory abnormality that precludes continuation of bosentan therapy
3. Pregnancy
4. AST and/or ALT values > 3 times the upper limit of normal range (ULN)
5. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C
6. Premature and permanent study drug discontinuation during the FUTURE 3 core study (AC-052-373)
7. Any major violation of the FUTURE 3 core study (AC-052-373) protocol.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2011-03-08 (Actual); Primary Completion 2014-08-13 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (3):
  - The Children's Hospital - Site 9102, Aurora, Colorado
  - Children's National Medical Center - Site 9104, Washington D.C., District of Columbia
  - Columbia University Medical Center Children's Hospital of New York Presbyterian - Site 9101, New York, New York
- Royal Children's Hospital Melbourne, Cardiology - Site 5001, Parkville, Australia
- The Republican Scientific-Practical Center "Cardiology" - Site 3001, Minsk, Belarus
- China (2):
  - Cardiovascular Institute and Fuwai Hospital, Beijing
  - Shanghai Children's Medical Center - Site 5102, Shanghai
- Fakultní nemocnice v Motole, dětské kardiocentrum - Site 3301, Prague, Czechia
- France (2):
  - Hopital Necker-Enfants Malades, Service de Cardiologie Pédiatrique - Site 2201, Paris
  - CHU de Toulouse - Hôpital des Enfants, Service de Cardiologie Pédiatrique - Site 2202, Toulouse
- Germany (3):
  - Deutsches Herzzentrum Kinderkardiologie - Site 1401, Berlin
  - Universitätsklinikum Bonn Abteilung für Kinderkardiologie - Site 1404, Bonn
  - Justus-Liebig-Universität Giessen, Kinderherzzentrum - Site 1403, Giessen
- Hungary (2):
  - Gottsegen György Országos Kardiológiai Intézet, Gyermekszív Központ, Gyermek Kardiológiai osztály - Site 3401, Budapest
  - Szegedi Tudományegyetem ÁOK Szent-Györgyi Albert Klinikai Központ, Gyermekgyógyászati Klinika és Gyermekegészségügyi Központ - Site 3402, Szeged
- CARE Hospitals, Cardiology Dep. Hyderabad - Site 5302, Hyderabad, India
- Schneider Children's Medical Center- Institute of pediatric cardiology - Site 7101, Petach Tikvah, Israel
- Italy (2):
  - Università Degli Studi di Padova - Dipartimento di Pediatria - Servizio di Cardiologia Pediatrica - Site 1501, Padua
  - Ospedale Pediatrico "Bambino Gesù" - Dipartimento Medico Chirurgico di Cardiologia Pediatrica - Site 1502, Rome
- Instituto Nacional de Cardiologia (INC) Ignacio Chavez - Site 8401, Mexico City, Mexico
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne Klinika Kardiologii Dziecięcej i Wad Wrodzonych Serca - Site 3604, Gdansk
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu Oddział Kardiologii Dziecięcej z pododdziałem Intensywnego Nadzoru Kardiologicznego - Site 3605, Wroclaw
- Russia (5):
  - RAMS Institution, Research Institute for complex issues of cardiovascular diseases, Siberian branch of the Russian Academy of Medical Sciences - Site 3805, Kemerovo
  - Scientific Center of Cardiovascular Surgery named after A.N.Bakulev of the RAMS - Site 3803, Moscow
  - Moscow Scientific Research Institute for Pediatrics and Childrens Surgery of Rosmedtechnologies - Site 3804, Moscow
  - Federal State Institution "Federal center of Heart, Blood and Endocrinology named after V.A.Almazov Rosmedtekhnologies" - Site 3802, Saint Petersberg
  - State Educational Institution of Higher Professional Education "Saint Petersburg State Pediatric Medical Academy of Roszdrav" - Site 3801, Saint Petersburg
- Serbia (2):
  - Univerzitetska dečja klinika, Služba za kardiologiju - Site 3901, Belgrade
  - Institut za zdravstvenu zaštitu majke i deteta Srbije "Dr Vukan Čupić", Služba za ispitivanje i lečenje bolesti srca i krvnih sudova - Site 3902, Belgrade
- South Africa (2):
  - Department of Paediatric Cardiology University of the Free State - Site 6001, Bloemfontein
  - Division of Paediatric Cardiology, Steve Biko Academic Hospital - Site 6002, Pretoria
- Spain (2):
  - Hospital Universitatario Vall d'Hebron, Neumologia - Site 1907, Barcelona
  - Hospital Universitario La Paz - Paediatric Cardiology Department - Site 1906, Madrid
- Ukraine (3):
  - Clinical Diagnostic Center - Pediatric Cardiovascular and ANES and Intensive Care Department - Site 4103, Dnipro
  - Gusak Ins Urgent and Recovery SUR AMS - Cardiovascular Rehabilitation Pediatric Department - Site 4101, Donetsk
  - Gover INS - Scientific Practical Cardiovascular Pediatric Center - MOH Ukraine - Site 4102, Kiev

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in this 1-year extension study were pediatric patients who completed the 6-month randomized open-label core study AC-052-373. In addition, patients were required to have tolerated study treatment during the FUTURE 3 core study and were considered by the investigator to benefit from continued bosentan treatment.
Pre-assignment Details: 64 patients were randomized in the FUTURE 3 core study, among whom 58 were enrolled in the FUTURE 3 extension study. Of the 58 participants in the FUTURE 3 extension study, a total of 10 participants entered the exceptional use treatment period (EUTP). Data for 3 participants in China after 19 Nov 2019 was not included in the report to meet the Human Genetic Resources Administration Office (HGRAO) requirements.
Groups:
- Bosentan 2mg/kg b.i.d.: Patients received 2 milligrams per kilogram (mg/kg) bosentan twice daily (b.i.d.) during the FUTURE 3 core study and continued with the same dose regimen during the extension study.
- Bosentan 2mg/kg t.i.d.: Patients received 2 mg/kg bosentan 3 times a day (t.i.d.) during the FUTURE 3 core study and continued with the same dose regimen during the extension study.
- Bosentan 2mg/kg b.i.d or t.i.d. During EUTP: Participants who entered the exceptional use treatment period (EUTP), continued receiving 2 mg/kg bosentan b.i.d or t.i.d up to Amendment B. After implementation of Amendment B, all participants received 2 mg/kg bosentan b.i.d.
Period: Core + Extension
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d. | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Started | 33 | 31 | 0
Enrolled in FUTURE 3 Extension | 31 | 27 | 0
Completed | 23 | 22 | 0
Not Completed | 10 | 9 | 0
Not completed — Adverse Event | 8 | 6 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Other (PAH not the main etiology of PH) | 0 | 2 | 0
Not completed — Other (administrative reason) | 1 | 0 | 0
Period: Exceptional Use Treatment Period
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d. | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Started | 0 | 0 | 10
Completed | 0 | 0 | 4
Not Completed | 0 | 0 | 6
Not completed — Administrative decision | 0 | 0 | 1
Not completed — Ongoing at the cut-off date of 19 Nov 2019 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d. | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at randomization in the FUTURE 3 core study (AC-052-373)
  years | 4.5 (3.35) | 5.2 (3.81) | 4.8 (3.57)
Age, Customized [Count of Participants; unit: Participants] — Number of subjects in each age category at randomization in the FUTURE 3 core study (AC-052-373)
  Participants
    Age Categories as per protocol: Infants and toddlers (28 days-23 months) | 10 | 11 | 21
    Age Categories as per protocol: Children (2-11 years) | 23 | 20 | 43
Sex: Female, Male [Count of Participants; unit: Participants] — Number of males and females randomized in the FUTURE 3 core study (AC-052-373)
  Participants
    Female | 18 | 10 | 28
    Male | 15 | 21 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race as per protocol: Caucasian/White | 25 | 23 | 48
  Race as per protocol: Black | 1 | 2 | 3
  Race as per protocol: Asian | 6 | 4 | 10
  Race as per protocol: Hispanic | 0 | 1 | 1
  Race as per protocol: Other | 1 | 1 | 2
Pulmonary Arterial Hypertension (PAH) etiology [Count of Participants; unit: Participants] — Children had a diagnosis of PAH belonging to one of the following categories: - Idiopathic PAH - Heritable PAH - Associated PAH persisting after complete repair of a congenital heart defect - PAH-congenital heart disease (PAH-CHD) associated with open shunts
  Participants
    Idiopathic | 14 | 15 | 29
    Heritable | 2 | 0 | 2
    Congenital heart disease | 6 | 2 | 8
    Associated PAH (i.e.,PAH after surgery for CHD) | 11 | 13 | 24
    Missing | 0 | 1 | 1
World Health Organization functional class (WHO FC) [Count of Participants; unit: Participants] — The World Health Organization (WHO) defines 4 classes to classify the functional status of patients with pulmonary hypertension: Class I (FC I): No limitation of physical activity; Class II (FC II): Slight limitation of physical activity; Class III (FC III): Marked limitation of physical activity; Class IV (FC IV): Inability to carry out any physical activity without symptoms.
  Participants
    FC I | 9 | 10 | 19
    FC II | 12 | 15 | 27
    FC III | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events (AEs) up to 7 Days After Permanent Study Drug Discontinuation
Description: This is the total number of subjects with at least one adverse event (serious or not serious) whether or not causally related to the study drug and presented cumulatively in the FUTURE 3 and FUTURE 3 Extension study. NOTE: FUTURE 3 extension study was exploratory and no primary efficacy and safety endpoints were defined in the protocol. So, this safety outcome measure was selected and reported as primary endpoint here.
Time Frame: Up to 62 weeks in average
Population: The analysis was performed on the Safety population analysis set, including all patients who received at least one dose of study treatment and evaluated according to the study treatment that they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d.
Number analyzed (Participants) | 33 | 31
Participants | 29 | 26

2. Other Pre Specified Outcome: Change From Baseline up to 12 Months of Study Treatment in the World Health Organization Functional Classification (WHO FC)
Description: The WHO FC indicates the severity of Pulmonary Arterial Hypertension: class I (none) to class IV (most severe). Changes from baseline to month 12 and month 18 of treatment with bosentan included: improvement (change from a higher to a lower FC), worsening (change from a lower to a higher FC) or no change/stable (same FC at baseline and at the post-baseline time point). Baseline was defined as the last valid assessment performed prior to first study drug intake in the FUTURE 3 core study.
Time Frame: At Month 12
Population: The intent to treat population was used. Where a missing visit score exists between two visits with scores, the missing score was imputed with the worse score of the non-missing scores; if the missing score was not between 2 visits with scores, it was replaced by the last non-missing score.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d.
Number analyzed (Participants) | 33 | 31
Participants
  Stable WHO FC | 22 | 25
  Improved WHO FC | 7 | 3
  Worsened WHO FC | 4 | 3

3. Other Pre Specified Outcome: Change From Baseline up to 18 Months of Study Treatment in the World Health Organization Functional Classification (WHO FC)
Description: as for outcome 2
Time Frame: At Month 18
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d.
Number analyzed (Participants) | 33 | 31
Participants
  Stable WHO FC | 25 | 25
  Improved WHO FC | 3 | 3
  Worsened WHO FC | 5 | 3

4. Other Pre Specified Outcome: Change From Baseline up to 12 Months of Study Treatment in the Global Clinical Impression Scale (GCIS)
Description: The GCIS is a scale used to rate the patient's current overall clinical condition ("Very Good", "Good", "Neither Good or Bad", "Bad", and "Very Bad"). Rating was performed independently by the physician and parents or legal representatives. Baseline was defined as the last valid assessment performed prior to first study drug intake in the FUTURE 3 core study.
Time Frame: At Month 12
Population: The intent to treat population was used for these analyses. No imputation method was used. Only patients with available results at the corresponding time point are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d.
Number analyzed (Participants) | 28 | 23
Participants
  Assessment by Physician: Stable | 16 | 16
  Assessment by Physician: Improved | 10 | 6
  Assessment by Physician: Worsened | 2 | 1
  Assessment by Parents/Legal representative: Stable | 16 | 12
  Assessment by Parents/Legal representative: Improved | 9 | 11
  Assessment by Parents/Legal representative: Worsened | 3 | 0

5. Other Pre Specified Outcome: Change From Baseline up to 18 Months of Study Treatment in the Global Clinical Impression Scale (GCIS)
Description: as for outcome 4
Time Frame: At Month 18
Population: The intent to treat population was used. No imputation method was used. Only patients with available results at the corresponding time point are including in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d.
Number analyzed (Participants) | 19 | 18
Participants
  Assessment by Physician: Stable | 9 | 12
  Assessment by Physician: Improved | 6 | 5
  Assessment by Physician: Worsened | 4 | 1
  Assessment by Parents/Legal representative: Stable | 8 | 7
  Assessment by Parents/Legal representative: Improved | 6 | 10
  Assessment by Parents/Legal representative: Worsened | 5 | 1

6. Other Pre Specified Outcome: Number of Patients With Pulmonary Arterial Hypertension (PAH) Worsening Components up to the Last Day of Treatment + 7 Days
Description: Number of patients with at least one PAH-worsening component (death, lung transplant, hospitalization due to PAH progression, initiation of new therapy for PAH, new/worsening right heart failure) reported cumulatively over FUTURE 3 core and extension study.
Time Frame: Up to 62 weeks in average
Population: The intent to treat population was used
Measure: Count of Participants; unit: Participants
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d.
Number analyzed (Participants) | 33 | 31
Participants
  At least one PAH-worsening event | 10 | 5
  No PAH-worsening event | 23 | 26

7. Other Pre Specified Outcome: Pulmonary Arterial Hypertension (PAH) Progression up to End of Treatment + 7 Days
Description: PAH progression was defined by time elapsed from the first study drug administration in the FUTURE core study to the day of the first occurrence of any of the following PAH worsening events: death, lung transplant, hospitalization due to PAH progression, initiation of new therapy for PAH or new / worsening right heart failure. Subjects without a PAH worsening event were censored at EOT + 7 days. PAH progression was estimated by Kaplan-Meier methodology and expressed by the percentage of participants free of events at different time points.
Time Frame: From baseline to Month 18
Population: These are the numbers of patients at risk at the time of study treatment initiation in the FUTURE 3 core study
Measure: Number (95% Confidence Interval); unit: Percentage of patients free of events
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d.
Number analyzed (Participants) | 33 | 31
Percentage of patients free of events
  Kaplan-Meier estimate at Month 12 | 74.9 [56.0 to 86.6] | 88.9 [69.4 to 96.3]
  Kaplan-Meier estimate at Month 18 | 68.2 [48.9 to 81.5] | 81.0 [60.1 to 91.7]
Statistical Analysis 1: Comparison: Bosentan 2mg/kg b.i.d. vs Bosentan 2mg/kg t.i.d; Post-hoc analysis: Cox proportional hazard regression univariate model with treatment as covariate (treatment-only univariate model); Test type: Other; Regression, Cox; Hazard Ratio (HR) = 1.438, 95% CI 2-sided [0.470 to 4.399]
Statistical Analysis 2: Comparison: Bosentan 2mg/kg b.i.d. vs Bosentan 2mg/kg t.i.d; Post-hoc analysis: Cox proportional hazard regression univariate model with WHO FC at baseline (FC III vs FC I/II) as covariate; Test type: Other; p = 0.0526, Regression, Cox — p-value <= 10% indicates that the covariate WHO FC at baseline is related to the time to PAH worsening
Statistical Analysis 3: Comparison: Bosentan 2mg/kg b.i.d. vs Bosentan 2mg/kg t.i.d; Post-hoc analysis: Treatment Hazard Ratio (HR) in the multivariate model with treatment and WHO FC at baseline as covariates; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 1.169, 95% CI [0.371 to 3.681]
Statistical Analysis 4: Comparison: Bosentan 2mg/kg b.i.d. vs Bosentan 2mg/kg t.i.d; Test of improvement in model fit from the univariate to the multivariate model with WHO FC at baseline as covariate; Test type: Superiority; p = 0.076, log(e) likelihood ratio — p-value <= 10% indicates an improvement in model fit

8. Other Pre Specified Outcome: Overall Survival
Description: Overall survival was defined as the time elapsed between the first study drug administration and death (any cause) up to end of study (Month 18 survival follow-up), regardless of whether the patient was on study treatment. Patients who died, regardless of the cause of death, were considered to have had an event. Patients last known to have been alive were censored on their date of last contact. Percentage of participants without death at different time points was estimated using Kaplan-Meier methodology.
Time Frame: From baseline to month 18
Population: These are the numbers of patients at risk at the time of study treatment initiation in the FUTURE 3 core study
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d.
Number analyzed (Participants) | 33 | 31
Percentage of participants
  Kaplan-Meier estimate at Month 12 | 81.8 [63.9 to 91.4] | 90.0 [72.1 to 96.7]
  Kaplan-Meier estimate at Month 18 | 75.8 [57.3 to 87.1] | 86.5 [68.0 to 94.7]
Statistical Analysis 1: Comparison: Bosentan 2mg/kg b.i.d. vs Bosentan 2mg/kg t.i.d; [analysis description as in outcome 7, analysis 1]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 1.935, 95% CI 2-sided [0.582 to 6.428]
Statistical Analysis 2: Comparison: Bosentan 2mg/kg b.i.d. vs Bosentan 2mg/kg t.i.d; [analysis description as in outcome 7, analysis 2]; Test type: Other; p = 0.0085, Regression, Cox; p-value <= 10% indicates that the covariate is related to the time to the time to death up to end-of-study
Statistical Analysis 3: Comparison: Bosentan 2mg/kg b.i.d. vs Bosentan 2mg/kg t.i.d; [analysis description as in outcome 7, analysis 3]; Test type: Other; Regression, Cox; Hazard Ratio (HR) = 1.487, 95% CI 2-sided [0.437 to 5.052]
Statistical Analysis 4: Comparison: Bosentan 2mg/kg b.i.d. vs Bosentan 2mg/kg t.i.d; Test of the improvement in model fit from the univariate to the multivariate model with WHO FC at baseline as covariate; Test type: Superiority; p = 0.014, log(e) likelihood ratio; p-value <= 10% indicates an improvement in model fit

9. Other Pre Specified Outcome: Exceptional Use Treatment Period (EUTP): Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) up to 7 Days After Permanent Discontinuation of Study Drug
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline.
Time Frame: Up to 7 days after discontinuation of study drug (up to 3 years and 4 months)
Population: Exceptional-use set included all patients who entered the EUTP. Due to change in study conduct, patients treated with bosentan t.i.d. switched to b.i.d. after local Amendment B to global protocol version 2 (17 March 2015 for Belarus and Ukraine, 1 April 2015 for China) and displaying summaries in the EUTP period by dose were not significant. Therefore, the results were reported combined for bosentan b.i.d./t.i.d.
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Number analyzed (Participants) | 10
percentage of participants | 80

10. Other Pre Specified Outcome: EUTP: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs) up to 7 Days After Permanent Discontinuation of Study Drug
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAE are defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 7 days after discontinuation of study drug (up to 3 years and 4 months)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Number analyzed (Participants) | 10
percentage of participants | 40

11. Other Pre Specified Outcome: EUTP: Percentage of Participants With AEs Leading to Premature Discontinuation of Study Drug
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Percentage of participants with AEs leading to premature discontinuation of study drug were reported.
Time Frame: Up to 3 years and 4 months
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Number analyzed (Participants) | 10
percentage of participants | 0

12. Other Pre Specified Outcome: EUTP: Percentage of Participants With SAEs From 7 up to 60 Days After Permanent Discontinuation of Study Drug
Description: A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From 7 up to 60 days after permanent discontinuation of study drug (up to 3 years and 4 months)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Number analyzed (Participants) | 10
percentage of participants | 0

13. Other Pre Specified Outcome: EUTP: Percentage of Participants With Deaths
Description: Percentage of participants with deaths were reported.
Time Frame: Up to 7 days after discontinuation of study drug (up to 3 years and 4 months)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Number analyzed (Participants) | 10
percentage of participants | 10

14. Other Pre Specified Outcome: EUTP: Percentage of Participants With Adverse Events of Special Interest (AESI)
Description: Percentage of participants with AESI including liver abnormalities and anemia were reported.
Time Frame: Up to 7 days after discontinuation of study drug (up to 3 years and 4 months)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Number analyzed (Participants) | 10
percentage of participants | 20

15. Other Pre Specified Outcome: EUTP: Percentage of Participants With Treatment-emergent Marked Laboratory Abnormalities up to 7 Days After Permanent Discontinuation of Study Drug
Description: Percentage of participants with treatment-emergent marked laboratory abnormalities were reported.
Time Frame: Up to 7 days after discontinuation of study drug (up to 3 years and 4 months)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Number analyzed (Participants) | 10
percentage of participants | 0

16. Other Pre Specified Outcome: EUTP: Percentage of Participants With Liver Function Abnormalities
Description: Percentage of participants with liver function abnormalities: Alanine aminotransferase (ALT) greater than (>)3*upper limit of normal (ULN), ALT/aspartate aminotransferase (AST) >3*ULN, ALT /AST >3*ULN and less than or equal to (<=) 5*ULN, ALT/AST >5*ULN and <=8*ULN, ALT/AST >8*ULN and ALT/AST >3*ULN, total bilirubin >2*ULN and alkaline phosphatase (ALP) <=2*ULN were reported.
Time Frame: Up to 7 days after discontinuation of study drug (up to 3 years and 4 months)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Number analyzed (Participants) | 10
percentage of participants | 0

17. Other Pre Specified Outcome: EUTP: Percentage of Participants With Any Time Occurrence of Hemoglobin <=10 Gram Per Deciliter (g/dL) and <=8g/dL Between Baseline and up to 7 Days After End of Treatment (EOT)
Description: Percentage of participants with any time occurrence of hemoglobin (Hgb) less than or equal to (<=) 10 g/dL and 8 g/dL between baseline and up to the last day of treatment + 7 days during EUTP were reported. Here "N" (number of subjects analyzed) signifies subjects who were evaluable for this outcome measure.
Time Frame: Baseline, up to 7 days after end of treatment (up to 3 years and 4 months)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
Number analyzed (Participants) | 9
percentage of participants
  Hgb <=10 g/dL | 22.2
  Hgb <=8 g/dL | 0

ADVERSE EVENTS:
Time Frame: From baseline up to end of treatment (and up to additional 60 days for serious adverse events and deaths), i.e. an average of 62 weeks and for EUTP: up to 7 days after discontinuation of study drug (approximately 3 years and 4 months)
Description: Adverse events are reported cumulatively for the FUTURE 3 core and extension studies
Groups:
- Bosentan 2mg/kg b.i.d.: 2 mg/kg bosentan was administered twice daily for a cumulative mean (± SD) duration of 64.1 ± 3.38 weeks (FUTURE 3 core + extension studies)
- Bosentan 2mg/kg t.i.d: 2 mg/kg bosentan was administered 3 times a day for a cumulative mean (± SD) duration of 60.4 ± 4.20 weeks (FUTURE 3 core + extension studies)
- Bosentan 2mg/kg b.i.d or t.i.d. During EUTP: Participants who entered the exceptional use treatment period (EUTP), continued receiving 2 mg/kg bosentan b.i.d or t.i.d up to Amendment B. After implementation of Amendment B, all participants received 2 mg/kg bosentan b.i.d. Due to change in study conduct, participants treated with bosentan t.i.d. switched to b.i.d. after local Amendment B to global protocol version 2 (17-03-2015 for Belarus and Ukraine, 1-04-2015 for China) and displaying summaries in the EUTP period by dose were not significant. Therefore, the data were combined for Bosentan b.i.d. and t.i.d.
Arm/Group | Bosentan 2mg/kg b.i.d. | Bosentan 2mg/kg t.i.d | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP
All-Cause Mortality (participants affected / at risk) | 8/33 | 4/31 | 1/10
Serious Adverse Events (participants affected / at risk) | 15/33 | 13/31 | 4/10
Other Adverse Events (participants affected / at risk) | 24/33 | 23/31 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bosentan 2mg/kg b.i.d. (N=33) | Bosentan 2mg/kg t.i.d (N=31) | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP (N=10)
ADENOIDAL HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIAL SEPTAL DEFECT REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC OPERATION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0)
CYANOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS ADENOVIRUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
METABOLIC DISORDER (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE WITH AURA (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
MUCOPOLYSACCHARIDOSIS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0) | 0 (0)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY HYPERTENSIVE CRISIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2)
PYREXIA (General disorders) | 0 (0) | 1 (2) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
SYNCOPE (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bosentan 2mg/kg b.i.d. (N=33) | Bosentan 2mg/kg t.i.d (N=31) | Bosentan 2mg/kg b.i.d or t.i.d. During EUTP (N=10)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (2) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 1 (1)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 6 (9) | 0 (0)
EAR INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 1 (1)
FLUSHING (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
LARYNGITIS (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 6 (16) | 5 (8) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 2 (5) | 1 (1) | 0 (0)
OTITIS MEDIA CHRONIC (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2)
PYREXIA (General disorders) | 5 (15) | 7 (15) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 1 (2) | 1 (2)
RHINITIS (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
TONSILLITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (22) | 13 (26) | 2 (2)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (6) | 3 (3) | 2 (2)
VOMITING (Gastrointestinal disorders) | 4 (5) | 6 (10) | 0 (0)
SPLENOMEGALY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
CYANOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
EXERCISE TOLERANCE DECREASED (General disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
VARICELLA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was uncontrolled and exploratory. The main purpose of exceptional use treatment period of FUTURE 3 extension was to provide participants with bosentan beyond 12-month treatment period of FUTURE 3 extension. Providing bosentan as a study treatment required monitoring safety on an individual participant-level. No formal hypothesis was formulated, therefore results were exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related article or abstract written independently by investigators must be submitted to Actelion for review at least 60 days prior to submission for publication or presentation.